CLINICAL TRIAL: NCT07097727
Title: Evaluation of the Role of Acetyl Cysteine in The Treatment of Ventilator Associated Pneumonia Induced by Carbapenem Resistance Klebsiella
Brief Title: Evaluation of the Role of Acetyl Cysteine in Ventilator Associated Pneumonia by Carbapenem Resistance Klebsiella
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Wessam Ibrahim Elfeky, Resident, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 36264MS321/9/23
Record Dates: First submitted 2025-07-11; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2023-10

CONDITIONS: Ventilator Associated Pneumonia ( VAP); Mechanical Ventilation
Keywords: Multi drug resistance; Ventilator-associated pneumonia; mechanical ventilation; carbapenem
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Acetylcysteine; Anti-Bacterial Agents; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acetyl cysteine 600 mg (Experimental): patients received acetyl cysteine 600 mg/ 12h IV in addition to antibiotics
  Interventions: Drug: acetyl cysteine 600 mg
- antibiotics and saline (Experimental): patients received only antibiotics and saline.
  Interventions: Drug: antibiotics and saline.

INTERVENTIONS:
Drug: acetyl cysteine 600 mg — patients received acetyl cysteine 600 mg/ 12h IV in addition to antibiotics
  Other Names: Group 1:intravenous infusion of acetyl cysteine 600 mg
  Arms: acetyl cysteine 600 mg
Drug: antibiotics and saline. — patients received only antibiotics and saline
  Other Names: Group 2 :antibiotics and intravenous infusion of 200 ml glucose 5%
  Arms: antibiotics and saline

SUMMARY:
The aim of the study is to evaluate the role of addition of Acetyl cysteine in the management of VAP induced by carbapenem resistant klebsiella. The primary outcome indicator is the change in modified clinical pulmonary infection score. The secondary outcome indicator is duration of mechanical ventilation.

DETAILED DESCRIPTION:
Ventilator-associated pneumonia remains the most common intensive care unit infection of patients on mechanical ventilation, and is associated with substantial morbidity/mortality, a longer hospital stays, and increased healthcare costs.

Multi drug resistance bacterial infection in Ventilator-associated pneumonia patients presents a global challenge due to its increasing morbidity and mortality. Multi drug resistance is defined as acquired nonsusceptibility to at least one agent in ≥ three antimicrobial categories according to the European Center for Disease Prevention and Control, The most common (80%) Ventilator-associated pneumonia pathogens were Pseudomonas aeruginosa, Acinetobacter baumannii, and Klebsiella pneumoniae.

Klebsiella pneumoniae is a common pathogen for community-and hospital-acquired infections, such as pneumonia, urinary tract infection, and bacteremia.

Infections due to Multi drug resistance Klebsiella species Were found to be associated with high mortality and hospital outbreaks. Carbapenem-resistant Klebsiella pneumoniae is among the bacteria that the World Health Organization gives critical priority to and poses the greatest threat to human health. According to China Antimicrobial Surveillance Network, carbapenem resistance in Klebsiella pneumoniae increased rapidly from 3% in 2005 to more than 25% in 2019. In case of new drugs unavailable or not active invitro, guidelines recommend combination of drugs active invitro (o polymyxins, aminoglycosides, tigecycline or Fosfomycin) with no recommendation for or against specific combinations.

In case of severe infections caused by Carbapenem-resistant Klebsiella carrying metallo-blactamases, guidelines recommend aztreonam and ceftazidimeavibactam combination therapy. Several studies demonstrated that acetyl Cysteine when added to antibacterial agent invitro, potentiates the antibacterial compound activities. The role of acetyl cystiene antioxidant and anti-inflammatory activities is being widely investigated in viral infections.

Since the mechanisms of acetyl cystiene effects in viral infections include its antioxidant and anti-inflammatory activities, they may also be beneficial in bacterial Multi drug resistance bacterial infections, The hypothesis of this study is that addition of acetyl cysteine to antibiotics in vivo could have a synergistic effect in Multi drug resistance bacterial infections and could help in decreasing high doses of antibiotics required, improving outcome and decrease hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are mechanically ventilated
* Age from 21 to 65
* Both sexes.

Exclusion Criteria:

* Patient guardians who refuse the consent • Hypersensitivity to acetyl Cysteine.
* Extrapulmonary infection.
* Cardiac patient with chronic heart failure
* Patient with lung diseases (tumors, tuberculosis, ,Chronic Obstructive Pulmonary Disease, Bronchiectasis and lung fibrosis)
* Severe immunosuppression (total leucocyte < 1000 mm3 or neutrophil < 500 cell/mm3.
* Patients on steroid or immunosuppressive drugs.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Improvement of clinical pulmonary infection score. | 14 days
  Improvement of clinical pulmonary infection score . score calculated in day 14 of treatment

SECONDARY OUTCOMES:
Duration of mechanical ventilation ventilation. | 14 days
  Duration of mechanical ventilation
mortality rate | 14 days
  Incidence of mortality

CONTACTS AND LOCATIONS:
Overall Officials: Wessam Elfeky, Resident, Principal Investigator — Tanta University
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: 6 months